CLINICAL TRIAL: NCT02661503
Title: HD21 for Advanced Stages Treatment Optimization Trial in the First-line Treatment of Advanced Stage Hodgkin Lymphoma; Comparison of 6 Cycles of Escalated BEACOPP With 6 Cycles of BrECADD
Brief Title: HD21 for Advanced Stages
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Prof., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1762; 2014-005130-55 (EudraCT Number)
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — Bleomycin; Etoposide; Doxorubicin; Cyclophosphamide; Vincristine; Procarbazine; Prednisone; Brentuximab Vedotin; Dacarbazine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BEACOPP (Active Comparator): 4 or 6 cycles of BEACOPP (21-day cycles) Bleomycin (B) Etoposide (E) Doxorubicin (A) Cyclophosphamide (C) Vincristine (O) Procarbazin (P) Prednisone (P). If FDG-PET is negative after two cycles patients will be given a total of four cycles. If FDG-PET is positive after two cycles patients will bev given a total of six cycles.
  Interventions: Drug: Bleomycin; Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Procarbazine; Drug: Prednisone
- BRECADD (Experimental): 4 or 6 cycles of BRECADD (21.day cycles) Brentuximab Vedotin (BR) Etoposide (E) Cyclophosphamide (C) Doxorubicin (A) Dacarbazine (D) Dexamethasone (D). If FDG-PET is negative after two cycles patients will be given a total of four cycles. If FDG-PET is positive after two cycles patients will be given a total of six cycles.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Brentuximab Vedotin; Drug: Dacarbazine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bleomycin
  Arms: BEACOPP
Drug: Etoposide
Drug: Doxorubicin
Drug: Cyclophosphamide
Drug: Vincristine
  Arms: BEACOPP
Drug: Procarbazine
  Arms: BEACOPP
Drug: Prednisone
  Arms: BEACOPP
Drug: Brentuximab Vedotin
  Arms: BRECADD
Drug: Dacarbazine
  Arms: BRECADD
Drug: Dexamethasone
  Arms: BRECADD

SUMMARY:
Primary objective of the trial is to demonstrate non-inferior efficacy of six cycles of BrECADD compared to six cycles of escalated BEACOPP, each followed by radiotherapy to PET-positive residual lesions ≥2.5 cm, in terms of progression free survival (efficacy objective).

If non-inferior efficacy can be shown, the co-primary objective is to further demonstrate reduced toxicity of the BrECADD treatment compared to the escalated BEACOPP treatment measured by treatment related morbidity (TRMorbidity objective).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven classical Hodgkin lymphoma
* First diagnosis, no previous treatment, 18 to 60 years of age
* Stage IIB with large mediastinal mass and/or extranodal lesions, stage III or IV

Exclusion Criteria:

* Composite lymphoma or nodular lymphocyte-predominant Hodgkin lymphoma
* Previous malignancy (exceptions: basalioma, carcinoma in situ of the cervix uteri, completely resected melanoma TNMpT1)
* Prior chemotherapy or radiotherapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1500 (Actual)
Dates: Start 2016-07; Primary Completion 2022-12 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 5 years
Treatment Related Morbidity | during 6 cycles of chemotherapy (21-day cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Borchmann, Prof., Principal Investigator — University of Cologne, I. Dept. of Medicine
Locations (1):
- University Hospital of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Ferdinandus J, Kaul H, Fossa A, Huttmann A, Keil F, Ko YD, Hitz F, Schwarz M, Trenker C, Kerkhoff A, Staib P, Wille K, Dresel I, Hahn D, Hertenstein B, Moosmann P, Mey U, Balabanov S, Armytage T, Roncolato F, Hellmuth JC, Hertzberg M, Kobe C, Klapper W, Baues C, Eich HT, Kreissl S, Fuchs M, Jablonski J, Schneider G, Tharmaseelan H, Eichenauer DA, von Tresckow B, Borchmann P, Brockelmann PJ. Positron Emission Tomography-Guided Brentuximab Vedotin, Etoposide, Cyclophosphamide, Doxorubicin, Dacarbazine, and Dexamethasone in Older Patients With Advanced-Stage Classic Hodgkin Lymphoma: A Prospective, Multicenter, Single-Arm, Phase II Cohort of the German Hodgkin Study Group HD21 Trial. J Clin Oncol. 2025 Sep 20;43(27):2974-2985. doi: 10.1200/JCO-25-00439. Epub 2025 Jul 17. PMID 40674676
- [Derived] Ferdinandus J, Schneider G, Moccia A, Greil R, Hertzberg M, Schaub V, Huttmann A, Keil F, Dierlamm J, Hanel M, Novak U, Meissner J, Hellmuth JC, Mathas S, Zijlstra JM, Fossa A, Viardot A, Hertenstein B, Martin S, Giri P, Kamper P, Molin D, Jablonski J, Damaschin C, Robertz AS, Rosenbrock J, Fuchs M, Borchmann P, Behringer K. Fertility in patients with advanced-stage classic Hodgkin lymphoma treated with BrECADD versus eBEACOPP: a secondary analysis of the multicentre, randomised, parallel, open-label, phase 3 HD21 trial. Lancet Oncol. 2025 Aug;26(8):1081-1090. doi: 10.1016/S1470-2045(25)00262-1. Epub 2025 Jul 10. PMID 40652943
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Borchmann P, Ferdinandus J, Schneider G, Moccia A, Greil R, Hertzberg M, Schaub V, Huttmann A, Keil F, Dierlamm J, Hanel M, Novak U, Meissner J, Zimmermann A, Mathas S, Zijlstra JM, Fossa A, Viardot A, Hertenstein B, Martin S, Giri P, Scholl S, Topp MS, Jung W, Vucinic V, Beck HJ, Kerkhoff A, Unger B, Rank A, Schroers R, Zum Buschenfelde CM, de Wit M, Trautmann-Grill K, Kamper P, Molin D, Kreissl S, Kaul H, von Tresckow B, Borchmann S, Behringer K, Fuchs M, Rosenwald A, Klapper W, Eich HT, Baues C, Zomas A, Hallek M, Dietlein M, Kobe C, Diehl V; German Hodgkin Study Group; Swiss Group for Clinical Cancer Research; Arbeitsgemeinschaft Medikamentose Tumortherapie; Nordic Lymphoma Group; Australasian Leukaemia and Lymphoma Group. Assessing the efficacy and tolerability of PET-guided BrECADD versus eBEACOPP in advanced-stage, classical Hodgkin lymphoma (HD21): a randomised, multicentre, parallel, open-label, phase 3 trial. Lancet. 2024 Jul 27;404(10450):341-352. doi: 10.1016/S0140-6736(24)01315-1. Epub 2024 Jul 3. PMID 38971175